CLINICAL TRIAL: NCT06888219
Title: REhabilitation of Dysphagia with ACupuncture and AuriculoTherapy in Non-communicative Patients with Severe Acquired Brain Injury (REDACT-Study): a Pilot Controlled Randomized Double Blinded Trial Study Protocol
Brief Title: Somatic and Ear Acupuncture for Dysphagia Rehabilitation and Decannulation After Severe Acquired Brain Injuries
Acronym: REDACT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REDACT
Record Dates: First submitted 2025-03-13; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-10

CONDITIONS: Brain Injury; Cognitive Impairment; Deglutition Disorder
Keywords: tracheostomy tube; acupuncture
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction; Deglutition Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture and Auriculotherapy (Experimental): Patients assigned to the intervention arm will receive conventional speech therapy rehabilitation (as in the control group) along with 2 or 3 weekly sessions of Acupuncture and Auriculotherapy, each lasting 20 minutes. The treatment will follow a protocol developed in collaboration with experienced acupuncture physicians and will involve the placement of approximately 10 somatic and auricular needles.
  Interventions: Other: Acupuncture and Auricolotherapy; Other: Conventional logopedic rehabilitation
- Conventional speech therapy rehabilitation (Active Comparator): Patients assigned to the control arm will undergo conventional speech therapy rehabilitation, which involves one hour per day of treatment, including restorative or passive compensatory interventions (e.g., modifications in food consistency and posture, passive exercises to improve swallowing structures) and the standard protocol for tracheal cannula weaning.
  Interventions: Other: Conventional logopedic rehabilitation

INTERVENTIONS:
Other: Acupuncture and Auricolotherapy — Based on the patient's condition and the physiology of traditional Chinese medicine, sterile disposable acupuncture needles will be placed on selected points:
  Auricular:
  * Esophagus point
  * Shen Men point
  * Palate area/ Throat point
  * II and III Trigeminal branches
  Somatic:
  * 17 Triple heater (if bruxisme)
  * 22 Conception Vessel
  * 23 Conception Vessel
  * 3 Small Intestine
  * Yin Tang (if apathy)
  * 3 Large Intestine (if xerostomy)
  * 36 and 44 Stomach
  Arms: Acupuncture and Auriculotherapy
Other: Conventional logopedic rehabilitation — Patients assigned to the control arm will undergo a total of 3 hours of speech and physiotherapy rehabilitation per day from Monday to Friday, and 1 hour on Saturday.
  Regarding speech therapy treatment, both restorative and compensatory interventions will be applied, based on the patient's clinical condition.
  Compensatory approaches include postural techniques (such as adopting a flexed head posture) and swallowing techniques (e.g., supraglottic swallowing, forced swallowing, the Mendelsohn maneuver), as well as modifying the consistency of liquids and food.
  Restorative methods involve swallowing exercises aimed at enhancing muscular strength, resistance training, and motor training of the oral structures involved in swallowing.

SUMMARY:
The goal of this interventional, randomized, controlled, double-blind pilot study is to assess the superiority of Acupuncture and Auriculotherapy, in addition to conventional speech therapy rehabilitation, for the treatment of dysphagia in patients with severe Acquired Brain Injury (sABI) of vascular etiology, who are tracheostomized and have severe cognitive impairment, classified as Level of Cognitive Functioning (LCF) <4 according to the LCF Scale.

The main questions this study aims to answer are:

* Does a treatment of 10 sessions of Acupuncture and Auriculotherapy, in addition to conventional speech therapy rehabilitation, help reduce dysphagia, as measured by clinical and instrumental scales, and shorten the time to decannulation after 4 weeks of treatment?
* Is the obtained result maintained 3 months after the end of the rehabilitation treatment?

Researchers will compare patients receiving conventional speech therapy rehabilitation with those also undergoing 10 sessions of Acupuncture and Auriculotherapy to determine whether this ancient Chinese technique can improve dysphagia and reduce time to decannulation in patients with vascular sABI and severe cognitive impairment.

Participants will be assigned to either the Intervention Group (Acupuncture and Auriculotherapy in addition to conventional rehabilitation) or the Control Group (conventional rehabilitation only). In both groups, conventional speech therapy rehabilitation will consist of 1 hour of treatment per day. The Intervention Group will undergo additional rehabilitation treatment using specific acupuncture and auriculotherapy points.

DETAILED DESCRIPTION:
On admission to the Intensive Rehabilitation Unit (IRU), patients with severe Acquired Brain Injury (sABI) often present with severe dysphagia (incidence up to 93%) and require a tracheal cannula (50-70%). During this intensive rehabilitation phase, the restoration of oral feeding and decannulation are two crucial and closely linked objectives. Studies have shown that the inability to manage saliva and dysphagia represents the main obstacle to decannulation, even in the long term.

Due to the extreme heterogeneity of patients with sABI and the lack of guidelines and consensus on the modalities and timing of dysphagia rehabilitation, swallowing rehabilitation still lacks standardization. Furthermore, most dysphagia rehabilitation techniques (both compensatory and restorative) require a certain degree of active patient collaboration, making them difficult to apply in sub-acute sABI patients.

In this context, acupuncture, which is already recommended by various international guidelines for conditions such as spasticity and pain, could be a valid therapeutic option. In fact, this technique has shown potential in reducing sialorrhea and muscular contractures in the oro-facial area, even in non-cooperative patients, such as those with a Disorder of Consciousness (DoC) or cognitive impairment.

This study aims to verify the effectiveness of Acupuncture and Auriculotherapy in the rehabilitation of dysphagia and tracheal cannula weaning in non-cooperative patients with sABI outcomes. The goal is to support the use of a safe, low-cost, bedside technique with no side effects, potentially applicable in all settings and during all rehabilitation phases.

The study will enroll 24 patients admitted to the IRU of the IRCCS-Fondazione Don Gnocchi of Florence for sABI of vascular etiology.

The baseline assessment (T0) at the time of study inclusion will involve the administration of clinical-instrumental scales to measure dysphagia severity:

* Mann Assessment of Swallowing Ability (MASA), assessed by the speech therapist
* Pooling Score, assessed by the phoniatrist using Fiberoptic Endoscopic Evaluation of Swallowing (FEES) A computerized randomization will assign patients to either the Intervention Group or the Control Group.

In both groups, conventional speech therapy rehabilitation will involve 1 hour per day of treatment, including restorative or passive compensatory interventions (e.g., modifications in food consistency and posture, passive exercises to improve swallowing structures) and the standard protocol for tracheal cannula weaning.

The Intervention Group will also undergo 2 or 3 weekly sessions of Acupuncture and Auriculotherapy, each lasting 20 minutes.

A follow-up clinical-instrumental assessment is scheduled:

At the end of 4 weeks of treatment (T1) At 3 months after T0 (T2)

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of severe Acquired Brain Injury with vascular etiology (ischemic or hemorrhagic), confirmed by Computerized Tomography or Magnetic Resonance Imaging.

Time between acute event and enrollment: 1 to 3 months. Age >18 years. Presence of a tracheal cannula upon admission to the Intensive Rehabilitation Unit.

Level of Cognitive Functioning (LCF) < or = 4. Informed consent signed by the patient's legal representative.

Exclusion Criteria:

Instability of general clinical conditions, including mechanical ventilation, sedation, sepsis or sub-emergent epileptic seizures.

Patients in Unresponsive Wakefulness Syndrome (UWS), according to the Coma Recovery Scale-Revised (CRS-R).

Known agoraphobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Significant difference measured by Mann Assessment of Swallowing Ability (MASA) Scale | From enrollment to the end of treatment at 4 weeks and at 3 months
  The Mann Assessment of Swallowing Ability (MASA) Scale consists of 26 items. The sum of the individual scores provides a total score that categorizes dysphagia and aspiration into four levels of severity.
  Dysphagia severity: The highest possible score is 200. 200-178: No abnormality detected 177-168: Mild dysphagia 167-139: Moderate dysphagia Below 138: Severe dysphagia (worst possible grade)
  Aspiration severity: The highest possible score is 200. 200-170: No abnormality detected 169-149: Mild aspiration 148-140: Moderate aspiration Below 140: Severe aspiration (worst possible grade)
Significant difference measured by Pooling Score, based on endoscopic landmarks and bedside parameters with relative values | From enrollment to the end of treatment at 4 weeks and at 3 months
  The Pooling Score is a clinical endoscopic evaluation used to assess the severity of swallowing disorders, considering excess residue in the pharynx and larynx.
  The score ranges from a minimum of 4 to a maximum of 11 and is calculated by summing the scores assigned to:
  Bolus location Amount of residue Ability to control residue/bolus pooling, assessed based on coughing, throat clearing (raclage), and the number of dry voluntary or reflex swallowing attempts (<2, 2-5, >5).

CONTACTS AND LOCATIONS:
Overall Officials: Bahia Hakiki, Principal Investigator — IRCCS-Fondazione Don Gnocchi
Locations (1):
- IRCCS-Fondazione Don Gnocchi, Florence, Italy

REFERENCES:
- [Background] Cohen DL, Roffe C, Beavan J, Blackett B, Fairfield CA, Hamdy S, Havard D, McFarlane M, McLauglin C, Randall M, Robson K, Scutt P, Smith C, Smithard D, Sprigg N, Warusevitane A, Watkins C, Woodhouse L, Bath PM. Post-stroke dysphagia: A review and design considerations for future trials. Int J Stroke. 2016 Jun;11(4):399-411. doi: 10.1177/1747493016639057. Epub 2016 Mar 22. PMID 27006423
- [Background] Garuti G, Reverberi C, Briganti A, Massobrio M, Lombardi F, Lusuardi M. Swallowing disorders in tracheostomised patients: a multidisciplinary/multiprofessional approach in decannulation protocols. Multidiscip Respir Med. 2014 Jun 20;9(1):36. doi: 10.1186/2049-6958-9-36. eCollection 2014. PMID 25006457
- [Background] Hakiki B, Draghi F, Pancani S, Portaccio E, Grippo A, Binazzi B, Tofani A, Scarpino M, Macchi C, Cecchi F. Decannulation After a Severe Acquired Brain Injury. Arch Phys Med Rehabil. 2020 Nov;101(11):1906-1913. doi: 10.1016/j.apmr.2020.05.004. Epub 2020 May 16. PMID 32428445
- [Background] Farneti D. Pooling score: an endoscopic model for evaluating severity of dysphagia. Acta Otorhinolaryngol Ital. 2008 Jun;28(3):135-40. PMID 18646575